CLINICAL TRIAL: NCT02490800
Title: An Open-label Phase 1/2a Study of Oral BAL101553 in Adult Patients With Advanced Solid Tumors and in Adult Patients With Recurrent or Progressive Glioblastoma or High-grade Glioma
Brief Title: Phase 1/2a Study of Oral BAL101553 in Adult Patients With Solid Tumors or Glioblastoma or High-grade Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDI-CS-002
Record Dates: First submitted 2015-06-25; First posted 2015-07-07 (Estimated); Results first posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Neoplasms
Keywords: Advanced solid tumors; Recurrent glioblastoma; High-grade glioma
MeSH Terms: conditions — Neoplasms; Glioblastoma; Glioma | interventions — lisavanbulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1 dose escalation portion (Experimental): Phase 1 dose escalation portion - an accelerated 3+3 titration design in patients with:
  1. advanced or recurrent solid tumors
  2. recurrent or progressive GBM / HGG
  Interventions: Drug: Lisavanbulin Phase 1 dose escalation portion
- Phase 2a dose expansion portion (Experimental): Phase 2a expansion portion (Simon's two-stage design) - Patients with recurrent and EB1-positive GBM
  Interventions: Drug: Lisavanbulin Phase 2a expansion portion

INTERVENTIONS:
Drug: Lisavanbulin Phase 1 dose escalation portion — Lisavanbulin hard capsules, containing 1 mg or 5 mg study drug, were given orally to fasted patients once daily in the dose range of 2 to 35 mg/day
  Other Names: BAL101553
  Arms: Phase 1 dose escalation portion
Drug: Lisavanbulin Phase 2a expansion portion — Recommended Phase 2 dose (RP2D) of 25 mg/day lisavanbulin hard capsules containing 5 mg study drug was administered once daily.
  Other Names: BAL101553
  Arms: Phase 2a dose expansion portion

SUMMARY:
First in human, open-label, dose escalation (Phase I) and expansion study (Phase 2a) of oral lisavanbulin (BAL101553) in adult patients with advanced solid tumors and adult patients with recurrent or progressive glioblastoma (GBM) or high-grade glioma (HGG).

DETAILED DESCRIPTION:
This was the first study of the oral formulation (hard capsules) of lisavanbulin. Lisavanbulin was administered once daily during each day of a 28-day treatment cycle to adults with advanced or recurrent solid tumors or recurrent or progressive GBM / HGG who had failed standard therapy, or for whom no effective standard therapy was available.

In Phase 1, the highest dose of lisavanbulin was determined that could safely be given to adults with advanced or recurrent solid tumors, recurrent or progressive GBM / HGG.

In Phase 2a, the tolerability and potential anticancer activity of oral lisavanbulin was assessed in patients with recurrent GBM whose tumor tissue tests positive for end-binding protein 1 (EB1). The study also measured pharmacokinetics.

ELIGIBILITY:
Main Inclusion Criteria:

1. Age ≥ 18 years
2. Patients who had in the Phase 1 portion either of the following:

   1. a histologically- or cytologically confirmed advanced or recurrent solid tumor, who failed standard therapy, or for whom no effective standard therapy was available to them
   2. histologically-confirmed GBM or HGG, with progressive or recurrent disease after prior radiotherapy, with or without chemotherapy. This also included patients with histologically-confirmed low-grade glioma who presented with unequivocal evidence by imaging of transformation to GBM / HGG

   Phase 2a dose expansion portion:

   Recurrent, histologically confirmed, glioblastoma with tumor tissue positive for EB1; eligible patients with de novo glioblastoma after prior radical chemo-radiotherapy or secondary glioblastoma after prior chemotherapy or radiotherapy.
3. Phase 1: Patients had to have measurable disease; according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1 for patients with advanced or recurrent solid tumors, and per radiological assessment in neuro-oncology (RANO) criteria for patients with recurrent or progressive GBM /HGG. Phase 2a: Patients had to be evaluable per RANO criteria.
4. Life expectancy ≥ 12 weeks
5. Acceptable organ and marrow function at baseline (protocol defined laboratory parameters)
6. Patients with advanced solid tumors had to have an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1 and patients with recurrent or progressive glioblastoma had to have an ECOG performance status ≤ 2

Main Exclusion Criteria:

1. Patients with advanced or recurrent solid tumors who had received chemotherapy, radiotherapy, immunotherapy, or investigational agents within 4 weeks (2 weeks for single fraction of palliative radiotherapy, 6 weeks for nitrosoureas or mitomycin C) prior to starting study drug or who had not recovered from side effects of prior therapies

   Patients with recurrent or progressive GBM / HGG who had: received radiotherapy within 6 weeks (Phase 1) or 12 weeks (Phase 2a), unless there was a new area of enhancement consistent with recurrent tumor outside the radiation field; received administration of prior anti-tumor chemotherapy within 4 weeks, or within 6 weeks for nitrosoureas; undergone surgical resection within 4 weeks (Phase 2a: 2 weeks) or a stereotactic biopsy/core biopsy within 1 week prior to starting study drug;
2. Patients who have had prior exposure to lisavanbulin
3. Inability to swallow oral medication
4. Increase in steroid dose in GBM or HGG patients within 5 days prior to first study-drug administration or requirement for > 6 mg/day dexamethasone or equivalent for symptom control.
5. Patients with gastrointestinal disease or those who have had a procedure that was expected to interfere with the oral absorption or tolerance of lisavanbulin
6. Symptomatic brain metastases or leptomeningeal disease, which was indicative of active disease, in patients with advanced or recurrent solid tumors.
7. Peripheral neuropathy ≥ CTCAE grade 2.
8. Uncontrolled intercurrent illness that would have unduly increased the risk of toxicity or limit compliance with study requirements
9. Systolic blood pressure (SBP) ≥ 160 mmHg or diastolic blood pressure (DBP) ≥ 100 mmHg at the screening visit.
10. Blood pressure (BP) combination treatment with more than two antihypertensive medications.
11. Women who were pregnant or breast-feeding. Men or women of reproductive potential who were not willing to apply effective birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-05-20 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Kaindl, MD, Study Director — Basilea Pharmaceutica International Ltd, Allschwil
Locations (13):
- UZ Leuven, Leuven, Belgium
- Germany (4):
  - Klinikum der Goethe-Universität Frankfurt, Frankfurt
  - Universitätsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Regensburg, Regensburg
  - Universitätsklinikum Tübingen, Tübingen
- Switzerland (4):
  - Universitätsspital Basel, Basel
  - Inselspital Universitätsspital Bern, Bern
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- United Kingdom (4):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - University College London NHS Foundation Trust, London
  - Sir Bobby Robson Cancer Trials Research Centre; Northern Centre for Cancer Care, Newcastle upon Tyne
  - Royal Marsden Hospital, Sutton

REFERENCES:
- [Derived] Lopez JS, Haefliger S, Plummer R, Clement PM, Jeffry Evans TR, Laubli H, Roth P, Kristeleit R, Brazil L, Tabatabai G, Wick A, Wunderlich B, Beebe K, Eisner JR, Lane H, Engelhardt M, Kaindl T, Hau P, Hundsberger T, Steinbach J. A phase 1/2a dose-finding study and biomarker assessment of oral lisavanbulin in patients with high-grade glioma or glioblastoma. Cell Rep Med. 2025 Jun 17;6(6):102165. doi: 10.1016/j.xcrm.2025.102165. PMID 40532659

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In the Phase 1 study, a total of 29 screening-failures occurred. Thus a total of 72 patients with advanced solid tumors, recurrent or progressive glioblastoma (GBM) or high-grade glioma (HGG) were enrolled in this Phase 1 and Phase 2a study.
Groups:
- Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day; Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day; Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day; Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day; Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day; Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day: Lisavanbulin hard capsules, containing 1 mg or 5 mg study drug, were given orally to fasted patients once daily
- Phase 2a Patients With Recurrent GBM: Lisavanbulin 25 mg/Day: The recommended Phase 2 dose (RP2D) of 25 mg/day lisavanbulin hard capsules containing 5 mg study drug was administered once daily.
Period: Overall Study
Arm/Group | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 2a Patients With Recurrent GBM: Lisavanbulin 25 mg/Day
Started | 3 | 3 | 3 | 7 | 7 | 3 | 4 | 3 | 7 | 3 | 8 | 3 | 18
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 7 | 7 | 3 | 4 | 3 | 7 | 3 | 8 | 3 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 2 | 3 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 3 | 3 | 3 | 4 | 4 | 1 | 4 | 3 | 6 | 2 | 7 | 1 | 10
Not completed — Patient enrolled in post-trial access | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Phase 2a Patients With Recurrent GBM: Lisavanbulin 25 mg/Day: RP2D of 25 mg/day lisavanbulin hard capsules containing 5 mg study drug was administered once daily
- Total: Total of all reporting groups
Arm/Group | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 2a Patients With Recurrent GBM: Lisavanbulin 25 mg/Day | Total
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 7 | 3 | 4 | 3 | 7 | 3 | 8 | 3 | 18 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.3 (21.94) | 66.7 (10.50) | 63.3 (6.51) | 61.0 (16.55) | 64.4 (7.00) | 65.7 (12.06) | 53.8 (9.95) | 53.7 (7.77) | 42.3 (9.62) | 45.3 (11.50) | 53.6 (9.78) | 51.3 (16.74) | 55.6 (10.43) | 55.7 (12.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5 | 6 | 0 | 2 | 2 | 3 | 2 | 2 | 1 | 3 | 31
  Male | 1 | 1 | 2 | 2 | 1 | 3 | 2 | 1 | 4 | 1 | 6 | 2 | 15 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 3 | 3 | 3 | 7 | 7 | 3 | 3 | 3 | 7 | 3 | 7 | 2 | 18 | 69
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Daily Oral Lisavanbulin
Description: First 28-day treatment cycle dose limiting toxicities (DLT) graded according to Common Terminology Criteria for Adverse Events (CTCAE) in the MTD-determining population in Phase 1 based on the number of participants with adverse effects as measure of tolerability at various dose levels
Time Frame: During first 28 day cycle
Population: MTD population: All patients from the safety set who met the following during the first 28-day treatment Cycle 1:
  * Received at least one dose of lisavanbulin and had experienced a DLT
  * Received at least 24 of the scheduled 28 doses for daily lisavanbulin administration, were not experiencing a DLT, had been observed for ≥ 28 days following the first dose, and had been evaluated for safety
Measure: Number; unit: mg
Groups:
- Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin: Lisavanbulin hard capsules, containing 1 mg or 5 mg study drug, were given orally to fasted patients once daily in the dose range of 2 to 30 mg/day
- Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin: Lisavanbulin hard capsules, containing 1 mg or 5 mg study drug, were given orally to fasted patients once daily in the dose range of 8 to 35 mg/day
Arm/Group | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin
Number analyzed (Participants) | 23 | 24
mg | 16 | 30

2. Primary Outcome: Phase 2a: Best Objective Response
Description: The best objective response was calculated as the proportion of patients responding (i.e., with a best observed objective response of complete or partial response) based on "radiological assessment in neuro-oncology (RANO)" criteria
Time Frame: Until the study discontinuation, on average 161 days (maximum of 381 days)
Population: The efficacy evaluable population (EEP) was the subset of the Full Analysis Population (FAP) who had at least one post baseline RANO assessment after having received at least 6 weeks of study treatment.
  For the primary endpoint, best objective response / objective response rate, the analysis was based on patients with measurable disease at baseline.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 2a Dose Expansion Portion: Phase 2a expansion portion (Simon's two-stage design) - Patients with recurrent and end-binding protein 1 (EB1)-positive GBM
  BAL101553 Phase 2a expansion portion: RP2D dose of 25 mg/day lisavanbulin hard capsules containing 5 mg study drug was administered once daily.
Arm/Group | Phase 2a Dose Expansion Portion
Number analyzed (Participants) | 9
Participants
  Complete response | 0
  Partial response | 1
  Stable disease | 4
  Progressive disease | 4

3. Primary Outcome: Phase 2a: Objective Response Rate (ORR)
Description: The ORR was calculated as the percentage of patients (rate) with complete and partial responses and its 95% Confidence Interval (CI) based on RANO criteria
Time Frame: Until the study discontinuation, on average 161 days (maximum of 381 days)
Population: Number of patients in EEP with measurable disease at baseline
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Phase 2a Dose Expansion Portion: Phase 2a expansion portion (Simon's two-stage design) - Patients with recurrent and EB1-positive GBM
  BAL101553 Phase 2a expansion portion: RP2D dose of 25 mg/day lisavanbulin hard capsules containing 5 mg study drug was administered once daily.
Arm/Group | Phase 2a Dose Expansion Portion
Number analyzed (Participants) | 9
Percentage of participants | 11.1 [0.3 to 48.2]

4. Secondary Outcome: Number of Patients With CTCAE Grade 3-4 TEAEs
Description: Number of patients experiencing treatment-emergent adverse events (TEAE) of CTCAE Grade 3 or 4
Time Frame: TEAEs were defined as all events occurring after lisavanbulin treatment began and up to 28 days after last study drug administration which corresponded to a maximum of 1653 days (4,5 years)
Population: Safety population: All patients who received at least one full or partial dose of lisavanbulin and had at least one post-baseline safety assessment
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 2a Patients With Recurrent GBM: Lisavanbulin 25 mg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 7 | 3 | 4 | 3 | 7 | 3 | 8 | 3 | 18
Participants
  Number of patients with only unrelated TEAEs of Grade 3-4 | 0 | 1 | 0 | 3 | 1 | 0 | 1 | 0 | 1 | 1 | 4 | 0 | 5
  Number of patients with related TEAEs of Grade 3-4 | 0 | 0 | 1 | 2 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Number of patients without TEAEs of Grade 3-4 | 3 | 2 | 2 | 2 | 2 | 1 | 3 | 3 | 6 | 2 | 4 | 2 | 10

5. Secondary Outcome: Cmax of Avanbulin (BAL27862)
Description: Pharmacokinetic parameter "Peak Plasma Concentration" Cmax of avanbulin Lisavanbulin (BAL101553) is the prodrug of avanbulin (BAL27862)
Time Frame: Plasma PK profiles were obtained on Cycle 1, Day 1 and on Cycle 2, Day 1 (pre-dose and from 0 up to 24 h post-dose) for all patients in the Phase 1 study who received lisavanbulin. For Phase 2 a study, PK parameters were obtained only on Cycle 1, Day 1
Population: The PK analysis set includes all patients who received at least one partial or complete dose of study drug (for the Phase 1 on Day 1 of Cycles 1 and 2, and for the Phase 2a only on Day 1 of Cycle 1) and had at least one post-baseline PK assessment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day; Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day; Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day: Lisavanbulin hard capsules, containing 1 mg or 5 mg study drug, were given orally to fasted patients once daily
- Phase 2a Cycle 1, Day 1 Patients With Recurrent GBM: Lisavanbulin 25 mg/Day: RP2D of 25 mg/day lisavanbulin hard capsules containing 5 mg study drug was administered once daily.
Arm/Group | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 2a Cycle 1, Day 1 Patients With Recurrent GBM: Lisavanbulin 25 mg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 7 | 5 | 7 | 3 | 3 | 4 | 3 | 3 | 3 | 7 | 4 | 3 | 2 | 8 | 6 | 3 | 1 | 18
ng/mL | 6.900 (0.580) | 9.800 (0.490) | 23.400 (0.440) | 40.880 (0.270) | 29.190 (0.490) | 44.270 (0.640) | 120.260 (0.490) | 109.560 (0.490) | 116.630 (0.580) | 147.730 (0.410) | 159.020 (0.080) | 35.260 (0.560) | 48.930 (0.910) | 75.130 (0.110) | 114.890 (0.430) | 64.110 (0.460) | 78.700 (0.640) | 103.950 (0.470) | 95.370 (0.110) | 146.500 (0.580) | 146.010 (0.340) | 159.100 (0.650) | 190.000 (NA) — Not evaluable | 98.210 (0.410)

6. Secondary Outcome: Tmax of Avanbulin (BAL27862)
Description: Pharmacokinetic parameter "Time to Peak Plasma Concentration" Tmax of avanbulin (BAL27862) Lisavanbulin (BAL101553) is the prodrug of avanbulin (BAL27862).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Median (Full Range); unit: Hours
Arm/Group | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 2a Cycle 1, Day 1 Patients With Recurrent GBM: Lisavanbulin 25 mg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 7 | 5 | 7 | 3 | 3 | 4 | 3 | 3 | 3 | 7 | 4 | 3 | 2 | 8 | 6 | 3 | 1 | 18
Hours | 2.0 [1.1 to 3.0] | 1.2 [1.0 to 2.0] | 1.1 [1.0 to 2.0] | 1.1 [1.0 to 2.0] | 3.0 [1.0 to 4.1] | 2.0 [1.1 to 4.0] | 1.1 [1.0 to 2.2] | 1.2 [1.0 to 2.2] | 1.0 [1.0 to 2.1] | 1.1 [1.0 to 2.1] | 2.0 [1.1 to 3.0] | 1.5 [1.0 to 2.2] | 1.0 [1.0 to 1.1] | 1.1 [0.8 to 2.0] | 1.1 [1.0 to 2.1] | 1.2 [0.6 to 2.2] | 1.1 [1.0 to 2.1] | 1.0 [1.0 to 2.0] | 2.0 [2.0 to 2.0] | 2.0 [0.5 to 3.0] | 2.0 [1.0 to 2.2] | 2.2 [2.1 to 3.1] | 1.0 [1.0 to 1.0] | 2.0 [0.6 to 3.0]

7. Secondary Outcome: AUC of Avanbulin (BAL27862)
Description: Pharmacokinetic parameter "Area under the plasma concentration versus time curve" AUC of avanbulin (BAL27862) Lisavanbulin (BAL101553) is the prodrug of avanbulin (BAL27862).
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Cycle 1, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 1 Cycle 2, Day 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 2a Cycle 1, Day 1 Patients With Recurrent GBM: Lisavanbulin 25 mg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 7 | 5 | 7 | 3 | 3 | 4 | 3 | 3 | 3 | 7 | 4 | 3 | 2 | 8 | 6 | 3 | 1 | 18
h*ng/mL | 34.040 (0.840) | 74.020 (0.830) | 180.060 (0.150) | 356.490 (0.160) | 258.460 (0.320) | 439.660 (0.620) | 823.980 (0.350) | 896.420 (0.540) | 1014.130 (0.650) | 1265.130 (0.410) | 1649.350 (0.250) | 230.800 (0.800) | 331.800 (1.760) | 692.230 (0.160) | 814.930 (0.460) | 344.540 (0.580) | 507.360 (0.740) | 575.060 (0.440) | 790.340 (0.110) | 1055.130 (0.250) | 1296.470 (0.370) | 1264.610 (0.320) | 1146.110 (NA) — Not evaluable | 713.710 (0.480)

8. Secondary Outcome: Phase 1: Best Objective Response
Description: The best objective response was calculated as the proportion of patients responding (i.e., with a best observed objective response of complete response (CR) or partial response (PR), according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria v1.1 for patients with advanced or recurrent solid tumors); and based on RANO criteria for patients with recurrent or progressive GBM / HGG
Time Frame: Until the end of treatment, on average 151 days (maximum of 1653 days), every other 28 day cycle
Population: Full analysis population (FAP): All patients who received at least one partial or complete dose of study drug, based on the intent-to-treat (ITT) principle
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 7 | 3 | 4 | 3 | 7 | 3 | 8 | 3
Participants
  Complete response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Partial response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Stable disease | 1 | 0 | 1 | 4 | 3 | 1 | 0 | 1 | 2 | 1 | 1 | 2
  Progressive disease | 2 | 3 | 2 | 2 | 4 | 2 | 4 | 2 | 5 | 1 | 5 | 1
  Missing | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

9. Secondary Outcome: Phase 1: Objective Response Rate (ORR)
Description: The ORR was calculated as the percentage of patients (rate) with complete and partial responses and its 95% CI based on RECIST criteria v1.1 for patients with advanced or recurrent solid tumors; and based on RANO criteria for patients with recurrent or progressive GBM / HGG
Time Frame: Until the study discontinuation, on average 151 days (maximum 1653 days), every other 28 day cycle
Population: FAP (Phase 1 portion of the study)
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Patients With Advanced or Recurrent Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day
Number analyzed (Participants) | 3 | 3 | 3 | 7 | 7 | 3 | 4 | 3 | 7 | 3 | 8 | 3
Percentage of patients | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 70.8] | 0 [0.0 to 41.0] | 0 [0.0 to 41.0] | 0 [0.0 to 70.8] | 0 [0.0 to 60.2] | 0 [0.0 to 70.8] | 0 [0.0 to 41.0] | 33.3 [0.8 to 90.6] | 12.5 [0.3 to 52.7] | 0 [0.0 to 70.8]

10. Secondary Outcome: Phase 2a: PFS
Description: PFS was defined as the interval between the date of drug administration and the earliest date of objective disease progression based on RANO criteria for patients with recurrent or progressive GBM / HGG. Patients who have not progressed or died at the end of the study were censored at the time of their latest objective tumor assessment.
Time Frame: 1 year
Population: PFS was summarized for the FAP and EEP
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Phase 2a Dose Expansion Portion (FAP); Phase 2a Dose Expansion Portion (EEP): Phase 2a expansion portion (Simon's two-stage design) - Patients with recurrent and EB1-positive GBM
  RP2D dose of 25 mg/day lisavanbulin hard capsules containing 5 mg study drug was administered once daily.
Arm/Group | Phase 2a Dose Expansion Portion (FAP) | Phase 2a Dose Expansion Portion (EEP)
Number analyzed (Participants) | 18 | 13
Months | 2.5 [1.4 to 7.5] | 3.5 [1.6 to NA] — Value(s) could not be evaluable due insufficient number of participants with events

11. Secondary Outcome: Phase 2a: PFS at 6 Months
Description: Percentage of patients without disease progression based on RANO criteria 6 months after the start of treatment. The values were determined using the Kaplan-Meier and Brookmeyer-Crowley methods.
Time Frame: 6 months
Population: FAP and EEP
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 2a Dose Expansion Portion (FAP) | Phase 2a Dose Expansion Portion (EEP)
Number analyzed (Participants) | 18 | 13
Percentage of participants | 31.3 [11.8 to 53.1] | 43.3 [16.3 to 67.9]

12. Secondary Outcome: Phase 2a: Overall Survival (OS) at 12 Months
Description: Percentage of patients alive 12 months after the start of treatment. The values were determined using the Kaplan-Meier and Brookmeyer-Crowley methods.
Time Frame: 1 year
Population: FAP and EEP
Measure: Median (95% Confidence Interval); unit: percentage of patients
Groups:
- Phase 2a Dose Expansion Portion (FAP); Phase 2a Dose Expansion Portion (EEP): Phase 2a expansion portion (Simon's two-stage design) - Patients with recurrent and EB1-positive GBM
  BAL101553 Phase 2a expansion portion: RP2D dose of 25 mg/day lisavanbulin hard capsules containing 5 mg study drug was administered once daily.
Arm/Group | Phase 2a Dose Expansion Portion (FAP) | Phase 2a Dose Expansion Portion (EEP)
Number analyzed (Participants) | 18 | 13
percentage of patients | 42.9 [15.9 to 67.8] | 55.6 [20.4 to 80.5]

ADVERSE EVENTS:
Time Frame: Treatment-emergent events occurring after lisavanbulin treatment began, up to 28 days after last study drug administration which corresponded to a maximum of 1653 days (4,5 years)
Groups:
- Phase 1 Patients Solid Tumors: Lisavanbulin 2 mg/Day; Phase 1 Patients With Solid Tumors: Lisavanbulin 4 mg/Day; Phase 1 Patients With Solid Tumors: Lisavanbulin 8 mg/Day; Phase 1 Patients With Solid Tumors: Lisavanbulin 16 mg/Day; Phase 1 Patients With Solid Tumors: Lisavanbulin 20 mg/Day; Phase 1 Patients With Solid Tumors: Lisavanbulin 30 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day; Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day: Lisavanbulin hard capsules, containing 1 mg or 5 mg study drug, were given orally to fasted patients once daily
Arm/Group | Phase 1 Patients Solid Tumors: Lisavanbulin 2 mg/Day | Phase 1 Patients With Solid Tumors: Lisavanbulin 4 mg/Day | Phase 1 Patients With Solid Tumors: Lisavanbulin 8 mg/Day | Phase 1 Patients With Solid Tumors: Lisavanbulin 16 mg/Day | Phase 1 Patients With Solid Tumors: Lisavanbulin 20 mg/Day | Phase 1 Patients With Solid Tumors: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day | Phase 2a Patients With Recurrent GBM: Lisavanbulin 25 mg/Day
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/7 | 0/7 | 0/3 | 0/4 | 0/3 | 1/7 | 0/3 | 1/8 | 0/3 | 7/18
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/3 | 0/3 | 4/7 | 5/7 | 1/3 | 0/4 | 0/3 | 2/7 | 1/3 | 4/8 | 2/3 | 8/18
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 6/7 | 7/7 | 3/3 | 4/4 | 3/3 | 5/7 | 3/3 | 7/8 | 3/3 | 18/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Patients Solid Tumors: Lisavanbulin 2 mg/Day (N=3) | Phase 1 Patients With Solid Tumors: Lisavanbulin 4 mg/Day (N=3) | Phase 1 Patients With Solid Tumors: Lisavanbulin 8 mg/Day (N=3) | Phase 1 Patients With Solid Tumors: Lisavanbulin 16 mg/Day (N=7) | Phase 1 Patients With Solid Tumors: Lisavanbulin 20 mg/Day (N=7) | Phase 1 Patients With Solid Tumors: Lisavanbulin 30 mg/Day (N=3) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day (N=4) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day (N=3) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day (N=7) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day (N=3) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day (N=8) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day (N=3) | Phase 2a Patients With Recurrent GBM: Lisavanbulin 25 mg/Day (N=18)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thalamic infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma prolapse (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 Patients Solid Tumors: Lisavanbulin 2 mg/Day (N=3) | Phase 1 Patients With Solid Tumors: Lisavanbulin 4 mg/Day (N=3) | Phase 1 Patients With Solid Tumors: Lisavanbulin 8 mg/Day (N=3) | Phase 1 Patients With Solid Tumors: Lisavanbulin 16 mg/Day (N=7) | Phase 1 Patients With Solid Tumors: Lisavanbulin 20 mg/Day (N=7) | Phase 1 Patients With Solid Tumors: Lisavanbulin 30 mg/Day (N=3) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 8 mg/Day (N=4) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 15 mg/Day (N=3) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 20 mg/Day (N=7) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 25 mg/Day (N=3) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 30 mg/Day (N=8) | Phase 1 Patients With Recurrent or Progressive GBM / HGG: Lisavanbulin 35 mg/Day (N=3) | Phase 2a Patients With Recurrent GBM: Lisavanbulin 25 mg/Day (N=18)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (5) | 0 (0) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 2 (2)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Neutrophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Brain oedema (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Hemianopia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Hyporesponsive to stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meralgia paraesthetica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neurologic neglect syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Partial seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 3 (6)
Sensory loss (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Cataract subcapsular (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Defaecation urgency (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 2 (2) | 0 (0) | 3 (5) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polyuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 2 (3) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (6)
Hypophagia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 0 (0) | 4 (4)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (8)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Early satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 8 (10)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Unevaluable event (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 6 (6)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychomotor retardation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnambulism (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT02490800/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-18): https://cdn.clinicaltrials.gov/large-docs/00/NCT02490800/SAP_001.pdf